CLINICAL TRIAL: NCT02195544
Title: Use of SYNVISC in Knee Osteoarthritis. Survey on Practice. "U.S.A.G.E Pratique"
Brief Title: Use of Synvisc® in Knee Osteoarthritis - Survey on Practice
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1139.5
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — hylan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Synvisc®
  Interventions: Drug: Synvisc®

INTERVENTIONS:
Drug: Synvisc®

SUMMARY:
Study of prescription methods in everyday medical practice, tolerance profile and effect of Synvisc® until six months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* not applicable

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: rheumatological practice
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 1998-10; Primary Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Change in clinical symptoms | up to 6 months
  assessed via questionnaire
Amount of medication consumed | up to 6 months
Patient satisfaction on a 4-point verbal rating scale | up to 6 months

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 6 months